CLINICAL TRIAL: NCT06826846
Title: Comparison of the Analgesic Effects of Continuous Serratus Posterior Superior Intercostal Plane Block With Catheter Versus Single-Shot Serratus Posterior Superior Intercostal Plane Block in Arthroscopic Shoulder Surgery
Brief Title: Comparison of the Analgesic Effects of Continuous Versus Single-Shot Serratus Posterior Superior Intercostal Plane Block in Arthroscopic Shoulder Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Goztepe Prof Dr Suleyman Yalcın City Hospital (Other)
Responsible Party: Principal Investigator, ILKER YALCIN, Anesthesiology and Reanimation Resident, M.D., Goztepe Prof Dr Suleyman Yalcın City Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: AOSPS001
Record Dates: First submitted 2025-02-10; First posted 2025-02-14 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-02

CONDITIONS: Arthroscopic Shoulder Surgery
Keywords: serratus posterior superior intercostal plane block; shoulder arthroscopy; regional anesthesia; plane block; postoperative pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Catheters

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1: This patient group will not undergo any regional block (No Intervention)
- Group 2: Patients who will receive a single-shot serratus posterior superior plane block (Active Comparator)
  Interventions: Other: Serratus posterior superior intercostal plane block (single-shot)
- Group 3: Patients who will receive a continuous SPSIB with catheter (Active Comparator)
  Interventions: Other: Serratus posterior superior intercostal plane block (catheter)

INTERVENTIONS:
Other: Serratus posterior superior intercostal plane block (single-shot) — 30 mL of 0.25% bupivacaine will be injected as single-shot block 20 mins prior to surgery
  Arms: Group 2: Patients who will receive a single-shot serratus posterior superior plane block
Other: Serratus posterior superior intercostal plane block (catheter) — In addition to administration of 30 mL of 0.25% bupivacaine prior to surgery, a catheter will be placed in the area to administer bolus of 1 mg/kg of 0.25% bupivacaine every 8 hours postoperatively.
  Arms: Group 3: Patients who will receive a continuous SPSIB with catheter

SUMMARY:
Patients undergoing arthroscopic shoulder surgery often experience moderate to severe postoperative pain. Various medical treatments are employed to provide analgesia for these patients. The advancement of regional anesthesia techniques has made possible to both reduce the use of narcotic analgesics and provide long-term pain management benefits.

The Serratus Posterior Superior Intercostal Plane Block (SPSIPB) was first described in 2023 by Serkan Tulgar et al. Cadaveric studies and dermatomal analyses in patients have demonstrated its ability to provide analgesia in the back, neck, shoulder, axilla, and lateral thoracic regions.

Even though patients undergoing shoulder surgery benefit from the block; once the duration of a single-shot block wears off, they may experience severe pain again. The aim of this study is to investigate the analgesic effects of a single-shot SPSIPB compared to continuous infusion provided by placing a catheter in this region.

The hypothesis of this study: In arthroscopic shoulder surgery, the continuous application of the serratus posterior superior intercostal plane block using a catheter will result in lower pain scores, reduced opioid consumption, and improved patient satisfaction compared to single-shot application.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18-80 years
* No bleeding diathesis
* Classified as ASA I-II-III

Exclusion Criteria:

* Patients who do not provide consent
* Patients with coagulopathy
* History of allergy or intoxication to local anesthetic agents
* Patients with advanced organ failure
* History of neuropathic disease
* Patients with mental retardation
* Presence of infection at the injection site
* Conditions in which regional anesthesia is contraindicated
* Pediatric patients and those over 80 years of age
* Pregnant patients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-09-15 (Actual); Study Completion 2025-10-10 (Actual)

PRIMARY OUTCOMES:
Postoperative Opioid Consumption | Postoperative 24 hours
  Patient-Controlled Analgesia (Tramadol)

SECONDARY OUTCOMES:
Postoperative Pain Scores | Postoperative 24 hours
  Tha pain will be assessed with Numeric Rating Scale at 0, 30 minutes, 1, 4, 8, 12, and 24 hours.
Patient Satisfaction (Likert scale) | Post surgery 24 hours
Postoperative Nausea and Vomiting Scale | 24 hours
Perioperative Remifentanyl Consumption | Perioperative assessment
Use of Rescue Analgesics in the Ward | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Senem Koruk, Study Director — Goztepe Prof Dr Suleyman Yalcın City Hospital
Locations (1):
- Goztepe Suleyman Yalcin City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No